CLINICAL TRIAL: NCT04778605
Title: Modulation of Endothelial Dysfonction Using Vitamin C in Septic Shock Patients
Acronym: MYTHICCS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP200301
Record Dates: First submitted 2021-02-26; First posted 2021-03-03 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-02

CONDITIONS: Septic Shock
Keywords: Endothelial dysfunction; Vitamin C; Septic shock; Microcirculatory effects; Hemodynamic effects
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with septic shock stabilized between H6 and H24 of treatment under noradrenaline.

SUMMARY:
Compare the microcirculatory reactivity before and after a 30-minute intravenous infusion of 40 mg/kg vitamin C and evaluate intra-individual variation of hemodynamic parameters between T0 and T1.

DETAILED DESCRIPTION:
This is a transversal study allowing to compare the microcirculatory reactivity before and after a 30-minute intravenous infusion of 40 mg/kg vitamin C.

Design:

• A monocentric, open-label, transversal study

Sample size :

30 patients

Assessement:

Between 6 hours and 24 hours after admission, the patient will be included after collection of the non opposition.

There will be two evaluation times: T0 before the start of vitamin C's perfusion, and T1: 1 hour after the end.

No interim analysis is planned. Analysis will be performed at the end of the study after data review and freezing of data base.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Septic shock patient, reanimated and stabilized defined as:

  * Patients with sepsis (suspected infection + 2 SOFA points) according to the latest international and the need to receive norepinephrine to maintain an average blood pressure above 65 mmHg
  * Patient supported for at least 6 hours, necessary for diagnostic management and hemodynamic optimization according to international standards and for less than 24 hours to limit confounding factors related to prolonged reanimation (sedation) and the empowerment of organ failures in general and vascular in particular. Hemodynamic stabilization will be defined as no increase in norepinephrine dosages

Exclusion Criteria:

* Pregnant or nursing women,
* Participation in another intervention research involving the human person or exclusion period following a previous research involving the human person
* Ward or curative patient
* Moribund patient
* Estimated life expectancy less than 1 month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: During septic shock, there are microcirculatory abnormalities, partly related to oxidative stress, which contribute to the pathophysiology of organ failures. We systematically supplement septic shock patients admitted in intensive care with vitamin C (ascorbic acid) because of the frequency of vitamin deficiencies in this population. Vitamin C having anti-oxidant properties, we hypothesized that Vitamin C's infusion could modulate microcirculatory endothelial reactivity in septic shock patients. This trial will allow us to include patients in stabilized septic shock between H6 and H24 of patient's care under norepinephrine.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-01-26 (Actual); Primary Completion 2021-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Compare the change in microcirculatory vascular reactivity before and after a 30-minute intravenous infusion of 40 mg / kg vitamin C. | 30 minutes
  Change (%) in microcirculatory vascular reactivity. T0 being measured just before the start of the vitamin C infusion. T1 being measured immediately after the 30-minute vitamin C infusion. The microcirculatory vascular reactivity will be evaluated using a cutaneous doppler laser coupled to an iontophoresis system. The doppler laser measures the skin perfusion on a sample of skin. A low intensity electric field is delivered for 12 seconds (3 times in a row at 1 minute interval) and allows local skin diffusion of an ionized solution of acetylcholine placed on the skin in a micro-sponge. It has been shown that this technique is very precise and that it is a very good reflection of endothelial function by measuring 3 parameters, the microcirculatory basal flow, the peak in response to acetylcholine and a more integrative index, the area under the curve with a standardized 10-minute recording. This local technique does not induce any side effects, it is very well tolerated.

SECONDARY OUTCOMES:
To study the hemodynamic effects of vitamin C on cardiac output, hemodynamic parameters: HR, BP, clinical perfusion parameters: marbling score, cutaneous re-coloring time. | 30 minutes
  Variation (%) in cardiac output between T0 and T1 (echocardiography) ((T1-T0) / T0x100).
  * Variation (%) of hemodynamic parameters between T0 and T1 ((T1-T0) / T0x100): Heart Rate, Blood Pressure, Cardiac output
  * Variation (%) of clinical perfusion parameters between T0 and T1 between T0 and T1: mottling score, skin recoloration time.
  All these parameters are routinely measured as part of the management of septic shock.

CONTACTS AND LOCATIONS:
Overall Officials: Hafid AIT-OUFELLA, Professor, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Intensive care department- Hôpital saint Antoine, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lavillegrand JR, Raia L, Urbina T, Hariri G, Gabarre P, Bonny V, Bige N, Baudel JL, Bruneel A, Dupre T, Guidet B, Maury E, Ait-Oufella H. Vitamin C improves microvascular reactivity and peripheral tissue perfusion in septic shock patients. Crit Care. 2022 Jan 21;26(1):25. doi: 10.1186/s13054-022-03891-8. PMID 35062987